CLINICAL TRIAL: NCT03511378
Title: An Open-label, Randomized, Comparative, Parallel Group Study to Assess the Immunogenicity of Lupin's Peg-filgrastim Versus Neulasta® as an Adjunct to Chemotherapy in Patients With Breast Cancer
Brief Title: Immunogenicity Assessment of Peg-filgrastim vs. Neulasta® as Adjunct to Chemotherapy in Patients With Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lupin Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LRP/PegGCSF/2016/004
Record Dates: First submitted 2018-03-20; First posted 2018-04-27 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
Keywords: Breast Carcinoma; Breast neoplasms; Breast Tumors; Cancer of Breast; Anti-Drug Antibodies (ADA); Immunogenicity
MeSH Terms: conditions — Breast Neoplasms | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lupin's Pegfilgrastim (Experimental): 6 mg, subcutaneous injection on day 2/3 of each 21 ± 3 day cycle. Number of cycles: 4.
  Interventions: Drug: Lupin's Pegfilgrastim
- Neulasta® (Experimental): 6 mg, subcutaneous injection on day 2/3 of each 21 ± 3 day cycle. Number of cycles: 4.
  Interventions: Drug: Neulasta®

INTERVENTIONS:
Drug: Lupin's Pegfilgrastim — Administration of Pegfilgrastim
  Other Names: INvestigational product
  Arms: Lupin's Pegfilgrastim
Drug: Neulasta® — Administration of Neulasta®
  Other Names: Reference
  Arms: Neulasta®

SUMMARY:
The purpose of this study is to compare the immunogenicity of Peg-filgrastim versus Neulasta® as an adjunct to chemotherapy in patients with breast cancer

DETAILED DESCRIPTION:
An open-label, randomized, comparative, parallel group study to assess the Immunogenicity of Lupin's Peg-filgrastim versus Neulasta® as an Adjunct to Chemotherapy in Patients with Breast Cancer

Primary Objective: To assess the immunogenicity of Lupin's Peg-filgrastim with Neulasta® in patients with breast cancer.

Secondary Objectives: To assess the safety of Lupin's Peg-filgrastim with Neulasta® in patients with breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able and willing to give written informed consent prior to any study related procedures
2. Ambulatory, female patients with an age ≥ 18 years
3. Patients with histologically or cytologically proven diagnosis of breast cancer who are eligible for neoadjuvant or adjuvant chemotherapy.
4. Patients who are planned and eligible to receive/ receiving myelosuppressive chemotherapy regimen that contains at least one chemotherapeutic agent from docetaxel/ paclitaxel / doxorubicin/ cyclophosphamide/ epirubicin
5. Patients who have not received any hematopoietic growth factors (e.g. G-CSF, PegGCSF, erythropoietin) or cytokines (e.g. interleukins, interferons) anytime in the past
6. Patients with baseline WBC ≥ LLN/ 3.5 x 109/L, ANC of ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L and hemoglobin ≥ 8.5 g/dL
7. Patients with ECOG Performance status of ≤ 2
8. Patient who have estimated life expectancy of more than six months
9. No evidences of hemorrhage

Exclusion Criteria:

1 Male patients

2. Hypersensitivity to any of the study drugs or its components like E.coli proteins or similar product

3. Patients weighing <45 Kg

4. Patients with myeloid malignancies and myelodysplasia or evidence of metastatic disease in bone marrow or brain

5. Patients currently receiving radiation therapy or have completed radiation therapy within 4 weeks before study entry or likely to receive radiotherapy during the study

6. Patients with prior bone marrow or stem cell transplantation

7. Patients with chronic use of oral corticosteroids (Except ≤ 20 mg/day dose of prednisolone/ equivalent steroids), immunotherapy, monoclonal antibody therapy and/or biological therapy or use of any other pegylated drug.

8. Patients with history of systemic antibiotic use within 72 hours prior to chemotherapy

9. Patients with any active infection which may require systemic antimicrobial therapy. Patients with inadequate hepatic and renal function [defined as Alkaline Phosphatase > 2.5 X Upper limits of normal (ULN), serum SGOT > 2.5 X ULN, SGPT > 2.5 X ULN, Total bilirubin > 1.5 X ULN and Creatinine > 1.5 X ULN of the reference range at the screening assessment]

10. Patients with seropositivity for HIV or HBV or HCV

11. Known cases of Sickle Cell Anemia

12. Patients with radiographic evidence of active pulmonary infections and/or recent history of pneumonia within 1 month of screening

13. Patients with clinically evident splenomegaly confirmed subsequently by ultrasonography

14. Patients with any other clinically significant disease(s) which, in the opinion of the investigator, could compromise the patient's involvement in the study or overall interpretation of the data. [for e.g. uncontrolled hematologic, renal, hepatic, endocrine, neurologic, psychiatric, metabolic, pulmonary, cardiovascular disease/impaired functioning or history of any autoimmune disease]

15. Patients who have participated in another therapeutic clinical study within the past 30 days prior to screening, or are likely to simultaneously participate in another therapeutic clinical study

16. Patients who are doubtful to comply with study procedures for mental, psychological or social reasons.

17. Women of child-bearing potential who are not willing to follow a reliable & effective contraceptive measure during the course of the study & at least 3 months after the last dose of study drug.

18. Pregnant and Breast feeding women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhananjay Bakhle, MD, Study Director — Lupin Limited
Locations (17):
- India (17):
  - M S Patel Cancer Centre,, Gokal, Anand
  - City Cancer Center, Vijayawada, Andhra Pradesh
  - Research & Development Department, HCG Cancer Center, Ahmedabad, Gujarat
  - Apple Hospital, Surat, Gujarat
  - Nirmal Hospital, Surat, Gujarat
  - Shree Himalaya Cancer Hospital & Research Institute,, Vadodara, Gujarat
  - Kailash Cancer Hospital & Research Center, Vadodara, Gujarat
  - Adhar health Institute, Hisar, Haryana
  - Sri Venketeshwara Hospital, Dept of Medical oncology, Bengaluru, Karnataka
  - Curie Manavata Cancer Centre, Mumbai, Maharashtra
  - Government Medical College & Hospital, Nagpur, Maharashtra
  - Sterling Hospital, Nigdi, Maharashtra
  - Bhaktivedanta Hospital & Research Institute, Thane, Maharashtra
  - Clinical Research Department, Bande, Nagpur
  - Acharya Tulsi Regional Cancer Treatment & Research Institute, Bīkaner, Rajahstan
  - Global Clinical Research Services Pvt Ltd., Hyderabad, Telangana
  - Apollo Gleneagles Hospitals, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The treatment group (Lupin pegfilgrastim or Neulasta®) for each patient during the study was determined according to the study randomization list. The treatment was assigned at the time of randomization, after confirming the patient's eligibility. Patients were randomized in a 1:1 ratio to receive either Lupin pegfilgrastim or Neulasta®.
Pre-assignment Details: All enrolled population included all screened patients who signed the informed consent. The randomized population included all randomized patients irrespective of whether patient received any study drug.
Groups:
- Lupin's Pegfilgrastim: 6 mg, subcutaneous injection on day 2 or 3 of each 21 ± 3 day cycle. Number of cycles: 4.
  Lupin's Pegfilgrastim: Administration of Pegfilgrastim
- Neulasta®: 6 mg, subcutaneous injection on day 2 or 3 of each 21 ± 3 day cycle. Number of cycles: 4.
  Neulasta®: Administration of Neulasta®
Period: Overall Study
Arm/Group | Lupin's Pegfilgrastim | Neulasta®
Started | 70 | 68
Completed | 67 | 66
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Patient not coming or schedule visit | 1 | 0

BASELINE CHARACTERISTICS:
Population: The enrolled patients were all middle-aged Asian females with a diagnosis of breast cancer.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lupin's Pegfilgrastim | Neulasta® | Total
Number analyzed (Participants) | 70 | 68 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (11.59) | 48.8 (8.73) | 51.2 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 68 | 138
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 70 | 68 | 138
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 70 | 68 | 138
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 70 | 68 | 138
ECOG Status at Screening [Count of Participants; unit: Participants] — The scale was developed by the Eastern Cooperative Oncology Group (ECOG). Grade 0: fully active. Grade 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature Grade 2: ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours Grade 3: capable of only limited self-care, confined to bed or chair more than 50% of waking hours Grade 4: completely disabled, cannot carry on any self-care, totally confined to bed or chair Grade 5: dead
  Participants
    Grade 0 | 20 | 16 | 36
    Grade 1 | 50 | 52 | 102
    Grade 2 | 0 | 0 | 0
    Grade 3 | 0 | 0 | 0
    Grade 4 | 0 | 0 | 0
    Grade 5 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Cumulative Incidence of Anti-pegfilgrastim Antibodies (Binding and Neutralizing) to Pegfilgrastim Between Treatment Groups at the End of Cycle 4 (Day 84).
Description: The difference in cumulative incidence of anti-pegfilgrastim antibodies (binding and neutralizing) (measured as difference in proportion of patients with antibodies) to Pegfilgrastim between study groups at the end of cycle 4 will be calculated. Those samples confirmed to be positive for binding antibodies were analyzed for presence of neutralizing antibodies to Pegfilgrastim.
Time Frame: End of cycle 4, Day 84
Population: Intention-to-treat analysis population
Measure: Number; unit: Proportion of patients with antibodies
Arm/Group | Lupin's Pegfilgrastim | Neulasta®
Number analyzed (Participants) | 69 | 68
Proportion of patients with antibodies | 0.0145 | 0.0441
Statistical Analysis 1: Comparison: Lupin's Pegfilgrastim vs Neulasta®; Analysis population : ITT; Test type: Non-Inferiority — Non-inferiority was assessed using a margin of -0.10; p = 0.007, Difference in proportion; Binomial proportion used to present difference in proportion in treatments; Difference in proportions = -0.0296, 95% CI 1-sided [lower limit -0.076]

2. Secondary Outcome: Comparison of Cumulative Incidence of Anti-peg Antibodies (Binding and Neutralizing) Between Treatment Groups at the End of Cycle 4 (Day 84).
Description: The presence of anti-peg antibodies (binding) (measured as difference in proportion of patients with antibodies) between treatment groups at the end of cycle 4 (Day 84) were compared and analysis for the ITT population
Time Frame: Day 84.
Population: Intention to treat population
Measure: Number; unit: Proportion of patients with antibodies
Arm/Group | Lupin's Pegfilgrastim | Neulasta®
Number analyzed (Participants) | 69 | 68
Proportion of patients with antibodies | 0.0145 | 0
Statistical Analysis 1: Comparison: Lupin's Pegfilgrastim vs Neulasta®; Analysis population: ITT; Test type: Non-Inferiority — Noninferiority is assessed using a margin of 10 percentage points; p < 0.001, Difference in proportion; Difference in proportions = 0.0145, 95% CI 1-sided [lower limit -0.0092] — Difference of proportion analysed with one sided 95% confidence interval

3. Secondary Outcome: Comparison of Incidence of Anti-pegfilgrastim Antibodies (Binding & Neutralizing) to Pegfilgrastim Between Treatment Groups on Day 10, Day 21, Day 42, Day 63 and Day 84
Description: Comparison of incidence of anti-pegfilgrastim antibodies (binding & neutralizing) (measured as difference in proportion of patients with antibodies) to pegfilgrastim between treatment groups on Day 10, Day 21, Day 42, Day 63, Day 84. Analysis population : ITT
Time Frame: Assessment at each study visit on Day 10, Day 21, Day 42, Day 63, Day 84
Population: The Intention-to-Treat (ITT) population included all patients who received at least one dose of study medication and subsequently provided immunogenicity variable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Lupin's Pegfilgrastim | Neulasta®
Number analyzed (Participants) | 69 | 68
Participants
  Day 10 | 1 | 0
  Day 21 | 0 | 1
  Day 42 | 1 | 1
  Day 63 | 0 | 1
  Day 84 (EOS) | 0 | 0

4. Secondary Outcome: Secondary Immunogenicity Endpoint
Description: Comparison of incidence of anti-peg antibodies (binding & neutralizing) (measured as difference in proportion of patients with antibodies) between treatment groups on Day 10, Day 21, Day 42, Day 63 and Day 84. Analysis population: ITT population
Time Frame: Day 10, Day 21, Day 42, Day 63 and Day 84.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Lupin's Pegfilgrastim | Neulasta®
Number analyzed (Participants) | 69 | 68
Participants
  Day 10 | 0 | 0
  Day 21 | 0 | 0
  Day 42 | 1 | 0
  Day 63 | 0 | 0
  Day 84 (EOS) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Any ongoing AE at the end of study visit were followed until the outcome was evident and resolved, clinically stabilized, or a plausible explanation had been found.
Arm/Group | Lupin's Pegfilgrastim | Neulasta®
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/70 | 2/68
Other Adverse Events (participants affected / at risk) | 57/70 | 56/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lupin's Pegfilgrastim (N=70) | Neulasta® (N=68)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lupin's Pegfilgrastim (N=70) | Neulasta® (N=68)
Vomiting (Gastrointestinal disorders) | 19 (24) | 20 (27)
Nausea (Gastrointestinal disorders) | 14 (16) | 18 (24)
Stomatitis (Gastrointestinal disorders) | 7 (9) | 5 (10)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 27 (28) | 22 (22)
Asthenia (General disorders) | 13 (17) | 15 (23)
Pain (General disorders) | 6 (7) | 8 (10)
Pyrexia (General disorders) | 3 (4) | 3 (4)
Mucosal inflammation (General disorders) | 3 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 6 (8)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 6 (8)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 9 (9)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Pyuria (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4)
Bacterial infection (Infections and infestations) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT03511378/Prot_SAP_000.pdf